CLINICAL TRIAL: NCT00549315
Title: Clinical Study of Thoracic Aortic Aneurysm Exclusion Using the VALIANT System
Brief Title: Clinical Study of Thoracic Aortic Aneurysm Exclusion
Acronym: Valiant
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Arizona Heart Institute (Other)
Responsible Party: Edward B. Diethrich, MD, Arizona Heart Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G020150
Record Dates: First submitted 2007-10-24; First posted 2007-10-25 (Estimated); Last update posted 2009-05-15 (Estimated); Status verified 2009-05

CONDITIONS: Thoracic Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Thoracic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Device: Valiant Endoluminal Stent-Graft Stent-Graft Balloon Catheter

INTERVENTIONS:
Device: Valiant Endoluminal Stent-Graft Stent-Graft Balloon Catheter — VALIANT stent-graft endoprosthesis is inserted by the Xcelerant Delivery System via a surgical cutdown (e.g., external iliac artery, femoral artery, common iliac artery conduit, etc.) approach. The insertion method depends on each patient's anatomy and is determined by the Clinical Investigator.

SUMMARY:
The Valiant stent-graft system is a flexible, implantable vascular stent-graft endoluminal device preloaded in a delivery system that is used to exclude thoracic aortic lesions (thoracic aneurysms, thoracic dissections, penetrating ulcers, traumatic transections and both traumatic and degenerative pseudoaneurysms.

DETAILED DESCRIPTION:
A vascular aneurysm is a permanent, localized dilatation of a blood vessel at least 1 1/2 to 2 times the normal vessel diameter. The aorta is the most frequent site for aneurysms, with approximately 10% of aortic aneurysms located above the renal arteries in the thoracic segment. Thoracic aortic aneurysms (TAAs) are less common than abdominal aorta, however, detection of TAAs is increasing, perhaps due to an aging population, increased diagnostic capability or an increase in prevalence.

Untreated thoracic aneurysms can be life-threatening. As many as 78% of untreated patients with TAA die within 5 years after diagnosis, most often from rupture of the aneurysm. Conventional surgical treatment, either tube graft placement or patch aortoplasty, is a high risk surgical procedure. Repair of the thoracic descending aorta is performed with a thoracotomy and cross-clamping of the aorta, with or without a shunt by-pass to maintain distal perfusion.

As an alternative to conventional surgery, a less invasive endovascular procedure has been developed that may be used to treat certain aneurysms. A collapsed stent-graft, a metal stent coupled with a fabric graft, is introduced into the vasculature, advanced to the size of the aneurysm, and deployed to span the aneurysm. The device creates a new aortic lumen, excluding the aneurysm sac from blood flow while maintaining flow within the stent-graft. This less invasive technique is designed to prevent or decrease the need for open surgery, to reduce the need for blood transfusion, to decrease the use of anesthetics and other drugs, and to speed recovery time. A reduction in intensive care and total hospital stay should result, leading to an increase quality of life following the procedure and a reduction in cost.

The primary objective of this investigational plan is to determine the safety of the Valiant endoluminal device when used to exclude thoracic lesions: true descending thoracic aortic aneurysms, dissections, penetrating ulcers, traumatic transections and traumatic and degenerative pseudoaneurysms from blood flow in high risk and low risk patients who are candidates for endoluminal repair.

Patients should be heparinized during the implant procedure (recommended activated clotting time is 200-300 seconds). During implantation of the Valiant endoluminal stent-graft, the pre-implant angiogram and CT scan are used together with (on-the-table) intravascular ultrasound (IVUS), digital subtraction angiography (DAS), roadmapping, and angiography for proper implant positioning. The Valiant endoluminal stent-graft endoprosthesis is inserted by delivery catheter and introducer sheath via a surgical cutdown (e.g., external iliac artery, femoral artery, common iliac artery conduit, etc.) approach. The introducer sheath and delivery catheter containing the stent-graft is inserted over a guidewire and advanced into the aorta and above the aneurysm. With the delivery catheter in the correct position, the introducer sheath is then withdrawn further until the stent-graft is completely deployed. A separate stent-graft balloon catheter system is provided with the device and may be used along the full length of the implanted device to model the springs against the vessel wall and to unravel possible wrinkles in the graft fabric. After deployment of the stent-graft, angiography is performed to verify implant position and to check for the presence of endoleaks.

Subjects will undergo an evaluation of the Valiant endoluminal stent-graft to determine the safety and efficacy of the device as indicated by the adverse event rate, and to determine the risk factors that are most predictive of a successful outcome when used to exclude thoracic aortic aneurysms that require suprarenal fixation in high risk and low risk patients. Follow-up will be completed at 1, 6, 12, 24, 36, 48, and 60 months. Subject evaluation at 1 month will include a Complete Physical Exam, Labs (BUN and Creatinine), and a Thoracic Spiral CT with and without IV contrast 2.5 mm. Subject evaluation at 6, 12, 24, 36, 48, and 60 months will include a Complete Physical Exam, Chest X-ray (AP, Lateral), Labs (BUN and Creatinine), and a Thoracic Spiral CT with and without IV contrast 2.5 mm.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥ 18 years of age.
* Subject is not pregnant or lactating. Females of child-bearing potential must practice a reliable method of contraception.
* Subject is diagnosed with one of the following conditions of the descending thoracic aorta. All conditions must be verified by diagnostic imaging [ultrasonography, computed tomography (CT), magnetic resonance imaging (MRI) or angiography].

  * A true (i.e., atherosclerotic) supraceliac aneurysm (fusiform or saccular type) with or without a co-existing aortic dissection or penetrating aortic ulcer;
  * Aortic dissection of DeBakey Type I or II (Stanford A, proximal) in the absence of an aneurysm; or
  * Penetrating aortic ulcer in the absence of an aneurysm; or
  * Traumatic transection; or
  * Pseudoaneurysm - traumatic or degenerative (i.e., one that does not involve all layers of the vessel and is not atherosclerotic in origin.
* Subject's anatomy is suitable for placement of the TALENT endoluminal stent-graft, with a distinct proximal aneurysm neck of 10 mm or more in length and a distal aneurysm neck of at least 10 mm.
* Subject has a TAA that is dilated to ≥ 5 cm in diameter, ≥ 1.5 times the diameter of the adjacent native/non-aneurysmal aorta, or is symptomatic.
* Subject has a proximal and distal aortic neck diameter ≥ 18 mm and ≤ 42 mm.
* Subject has an arterial access site, either peripherally or via infrarenal abdominal aorta that is adequate for introduction of the stent-graft delivery system.
* Subject has signed the informed consent.
* Subject will be available for the periodic follow-up (surveillance) after the procedure.
* Aortic.

Exclusion Criteria:

* Subject has TAA with less than 10 mm proximal fixation length.
* Subject has an aneurysm that would require exclusion by the stent-graft of the segment of the aorta that gives rise to dominant spinal cord/intercostal arteries.
* Subject has a lesion that prevents delivery or expansion of the device.
* Subject has systemic infection, or is suspected of having systemic infection.
* Subject has a known mycotic aneurysm.
* Subject is not available or is not willing to come back for periodic follow-up (surveillance) after the procedure.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2002-10; Primary Completion 2012-09 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Determine the proportion in whom successful implantation is achieved, as indicated by aneurysm exclusion and graft patency. | At implant, time of discharge, and 1, 6, and 12 months.

SECONDARY OUTCOMES:
Determine the proportion of patients who experience adverse events. | During and after implantation.
Determine the proportion of patients who experience comorbidities and overall mortality rates. | During and after implantation.

CONTACTS AND LOCATIONS:
Overall Officials: Edward B Diethrich, M.D., Principal Investigator — Arizona Heart Institute
Locations (1):
- Arizona Heart Institute, Phoenix, Arizona, United States

REFERENCES:
- [Background] Coselli JS, S Buket, and ES Crawford. 1996. Thoracic aortic aneurysms. In: Haimovicis Vascular Surgery, 4th ed, H Haimovici, E Ascer, LH Hollier, DE Strandness, and JB Towne, eds. Blackwell Science, chapter 57.
- [Background] Coselli JS and SA LeMaire. 1995. Diseases of the thoracic aorta. In: Current Diagnosis and Treatment in Vascular Surgery, 1st ed, RH Dean, JST Yao, and DC Brewster, eds. Appleton & Lange, Norwalk, CT, chapter 11.
- [Background] Dake MD, Miller DC, Semba CP, Mitchell RS, Walker PJ, Liddell RP. Transluminal placement of endovascular stent-grafts for the treatment of descending thoracic aortic aneurysms. N Engl J Med. 1994 Dec 29;331(26):1729-34. doi: 10.1056/NEJM199412293312601. PMID 7984192
- [Background] Mitchell RS, Miller DC, Dake MD. Stent-graft repair of thoracic aortic aneurysms. Semin Vasc Surg. 1997 Dec;10(4):257-71. PMID 9431597
- [Background] Moreno-Cabral CE, Miller DC, Mitchell RS, Stinson EB, Oyer PE, Jamieson SW, Shumway NE. Degenerative and atherosclerotic aneurysms of the thoracic aorta. Determinants of early and late surgical outcome. J Thorac Cardiovasc Surg. 1984 Dec;88(6):1020-32. PMID 6503314
- [Background] Najafi H. Thoracic aortic aneurysm: evaluation and surgical management. Compr Ther. 1994;20(5):282-8. No abstract available. PMID 8045085
- [Background] Pressler V, McNamara JJ. Thoracic aortic aneurysm: natural history and treatment. J Thorac Cardiovasc Surg. 1980 Apr;79(4):489-98. No abstract available. PMID 7359927
- [Background] Skeens JL and MD Dake. 1997. Thoracic aortic aneurysm stent-grafts. Eighth Complex Peripheral Angioplasty Course. Paris, May 20-23, 1997, pp. 289-295.
- [Background] Nienaber CA, Fattori R, Lund G, Dieckmann C, Wolf W, von Kodolitsch Y, Nicolas V, Pierangeli A. Nonsurgical reconstruction of thoracic aortic dissection by stent-graft placement. N Engl J Med. 1999 May 20;340(20):1539-45. doi: 10.1056/NEJM199905203402003. PMID 10332015
- [Background] White RA, Donayre CE, Walot I, Lippmann M, Woody J, Lee J, Kim N, Kopchok GE, Fogarty TJ. Endovascular exclusion of descending thoracic aortic aneurysms and chronic dissections: Initial clinical results with the AneuRx device. J Vasc Surg. 2001 May;33(5):927-34. doi: 10.1067/mva.2001.114998. PMID 11331830